CLINICAL TRIAL: NCT04535687
Title: Fluzoparib in Patients With Metastatic Non-clear Cell Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCC-MUL-IIT-FZPL
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Fluzoparib alone
  Interventions: Drug: Fluzoparib

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib

SUMMARY:
This trial aims to prospectively assess the safety and efficiency of Fluzoparib in metastatic non-clear cell renal cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years of age or older
* Histological proof of metastatic non-clear cell renal cell carcinoma (AJCC Stage IV)，Must have measurable disease as defined by RECIST 1.1 criteria
* Somatic or germline mutation in homologous recombination gene from tissue, saliva or blood-based genetic test
* At least one prior treatment with a Tyrosine Kinase Inhibitor，the progress of soft tissue lesions need to be consistent with RECIST1.1
* Any number of prior systemic therapies is allowed (cytokine, anti-angiogenic, mTOR, immune checkpoint blockage or clinical trial)
* Participants must have a life expectancy ≥ 3 months
* ECOG PS ≤ 1
* Participants must have normal organ and bone marrow function measured within 14 days prior to administration of study treatment as defined below：
* Hemoglobin ≥ 100 g/L
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional ULN
* Blood Urea Nitrogen（BUN）/Creatinine(Cr)≤ 1.5 x institutional ULN
* Appropriate measures should be taken for contraception for women in childbearing period and man with reproductive capacity
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Other malignancy unless curatively treated with no evidence of disease for ≥ 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma. Patients with a history of localized triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy > 3 years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with symptomatic uncontrolled brain metastases. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Judged by investigator, the subjects had other factors that could lead to the termination of the study such as with other serious disease (including mental illness) need to merge treatment, serious abnormal laboratory values, family and social factors maybe affect the safety or data collection
* Breast feeding women
* Use of any prohibited concomitant medications within the prior 2 weeks
* Involvement in the planning and/or conduct of the study
* Participation in another clinical study with an investigational product during the last 4 weeks
* Patients receiving any systemic chemotherapy or radiotherapy within 4 weeks prior to study treatment
* Any previous treatment with PARP inhibitor, including fluzoparib
* Subjects Have failed to control the heart of the clinical symptoms or disease, such as: (1) the NYHA class II or worse heart failure；(2)unstable angina pectoris；(3)myocardial infarction occurred within 1 year；(4) Patients with clinically significant ventricular or ventricular arrhythmia requiring clinical intervention; (5) QTc≥470ms
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting fluzoparib is 2 weeks
* Concomitant use of known strong CYP3A inducers (e.g. phenobarbital, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting fluzoparib is 5 weeks for phenobarbital or enzalutamide and 3 weeks for other agents
* Adverse events caused by previously accepted treatment（except hair loss ） have not recovered (grade 1 or baseline level) or less
* Patients with myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery
* Unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Poor medical risk due to a serious, uncontrolled non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled uncontrolled major seizure disorder, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan
* Congenital or acquired immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV)
* Known hypersensitivity to fluzoparib or any of the excipients of the product
* Known active hepatitis (i.e. Hepatitis B：HBsAg positive，HBV DNA≥2000IU/ml or copy number≥10000/ml；Hepatitis B：HCV antibodies positive，copy number≥institutional ULN)
* Uncontrolled hypertension, defined as systolic blood pressure (BP) >= 150 millimeters of mercury (mmHg) or diastolic BP >= 100 mmHg with or without antihypertensive dication
* Packed red blood cells and/or platelet transfusions within the last 28 days prior to study entry
* Abnormal coagulation function（INR>2.0，PT>16s），hemorrhagic tendency or undergoing thrombolytic or anticoagulant therapy. The patient can receive low dose aspirin, low molecular weight heparin for precausion

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
objective response rate（ORR） | three months
  the proportion of patients with CR, PR, and SD in the group（RECIST1.1）

SECONDARY OUTCOMES:
radiographic progression free survival（rPFS） | six months
  the time frame from the first day of fluzoparib to the date of radiographic confirmed progressive disease or death which one occurrs first
overall survival（OS） | eighteen months
  the time frame from the first day of fluzoparib to the date of death the time frame from the first day of apatinib to the date of death the time frame from the first day of apatinib to the date of death the time frame from the first day of apatinib to the date of death the time frame from the first day of apatinib to the date of death
time to progression（TTP） | six months
  the time frame from the first day of fluzoparib to the date of confirmed progressive
AE | 2 years
  Number of Adverse Events, Grade 3 or higher as defined by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, Phd, Study Chair — Department of Urology, Drum Tower Hospital, Medical School of Nanjing University
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China